CLINICAL TRIAL: NCT04914689
Title: External Focus of Attention Feedback to Reduce Risk of Non-contact ACL Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Responsible Party: Principal Investigator, Abbey Thomas, PhD, Assistant Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-0283
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal focus of attention feedback (Active Comparator): Participants will complete 12 sessions over 3 weeks receiving visual feedback in a mirror of their movement patterns.
  Interventions: Other: Internal focus of attention feedback
- Visual external focus of attention feedback (Experimental): Participants will complete 12 sessions over 3 weeks receiving visual feedback of their movement patterns from a laser.
  Interventions: Other: Visual internal focus of attention feedback
- Auditory external focus of attention feedback (Experimental): Participants will complete 12 sessions over 3 weeks receiving auditory feedback of their movement patterns.
  Interventions: Other: Auditory external focus of attention feedback

INTERVENTIONS:
Other: Internal focus of attention feedback — Participants will complete 12 sessions over a 3-week period of functional movement retraining while receiving mirror feedback. Participants will be instructed to perform each functional task in a manner that keeps their knee in line with their toes.
  Arms: Internal focus of attention feedback
Other: Visual internal focus of attention feedback — Participants will complete 12 sessions over a 3-week period of functional movement retraining while receiving visual feedback via laser. Participants will be instructed to perform each functional task in a manner that does causes the laser to move up and down but not side-to-side.
  Arms: Visual external focus of attention feedback
Other: Auditory external focus of attention feedback — Participants will complete 12 sessions over a 3-week period of functional movement retraining while receiving auditory feedback. Participants will be instructed to perform each functional task in a manner that does not cause the auditory tool to elicit a noise.
  Arms: Auditory external focus of attention feedback

SUMMARY:
Knee injuries, especially those to the ACL, are common among physically active people. Preventing these injuries from happening is critical to limiting the long-term pain, disability, and arthritis associated with these injuries. Our study is going to examine new ways to provide feedback about the way people move to determine if these are better at modifying movement patterns to prevent injury than current standard treatments. If you participate, you will be asked to undergo a movement analysis in a research laboratory while you perform tasks such as landing from a box and running and cutting. After this initial assessment, you will be randomly allocated to one of 3 treatment groups. Each treatment group will perform 4 weeks (3x/week) of exercises to change the way people land from a jump. Participants will then report for follow-up movement analysis testing 1- and 4-weeks after completing the intervention.

DETAILED DESCRIPTION:
Despite the popularity of injury prevention programs, anterior cruciate ligament (ACL) injuries continue to occur at a rate of 250,000 per year in the United States. It is believed that 75% of these injuries are preventable, thus alternative strategies to reduce the risk of injury are necessary. One reason current prevention strategies are not wholly successful may be their reliance on internal focus of attention (InFOCUS) feedback, which constrains movement and increases injury risk. Our project will examine an alternative approach, testing two different modes of external focus of attention (ExFOCUS) feedback to remove constrains on the way people move to reduce injury risk. We will also examine cortical activity to determine if there are differences in neuroplasticity that occur following each form of feedback to better understand how each works. Collectively, the knowledge gained from this study will inform the development of programs to reduce injury risk.

Specific Aim 1: Determine ExFOCUS's ability to reduce the risk of noncontact ACL injury by retaining improved biomechanics compared to InFOCUS. Hypothesis 1.1: the combined auditory and visual ExFOCUS groups will demonstrate greater improvements in biomechanics and will retain these improvements 1 month after cessation of the intervention.

Specific Aim 2: Determine differences in the ability of the two modes (visual and auditory) of ExFOCUS to change biomechanics. Hypothesis 2.1: Auditory ExFOCUS feedback will elicit superior results compared to visual ExFOCUS feedback immediately following the intervention. Specific Aim 3: To quantify differences in cortical activity following external focus of attention and internal focus of attention feedback. Hypothesis 3.1: External focus of attention feedback will increase cortical activity in both groups while there will be no changes in cortical activity during internal focus of attention feedback Hypothesis 3.2: Auditory feedback will elicit greater changes in auditory regions of the brain, while visual feedback will elicit greater changes in regions of the brain responsible for processing visual information.

ELIGIBILITY:
Inclusion Criteria:

* exercise 30+ minutes 3+ days/week

Exclusion Criteria:

* Body mass index >40 kg/m2
* History of lower extremity fracture or surgery to either limb
* History of ACL tear, meniscus, or collateral ligament injury at the knee to either limb
* History of ankle sprains to either limb
* History of musculoskeletal injury sustained in the 6 months prior to enrollment
* History of concussion or neurological disorders that may influence electroencephalography activity
* Visual or hearing impairments that would limit receiving the appropriate feedback
* Inability to comprehend and repeat back directions in English
* Current smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in lower extremity biomechanics during landing. | 1-week post-intervention, 4-weeks post-intervention
  Hip and knee angles and loads measured via 3D biomechanics
Differences in biomechanical changes between visual and auditory external focus of attention feedback. | 1-week post-intervention, 4-weeks post-intervention
  Hip and knee angles and loads measured via 3D biomechanics

SECONDARY OUTCOMES:
Changes from baseline in cortical activity during landing | 1-week post-intervention, 4-weeks post-intervention
  Electroencephalography recording of cortical activity during landing

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No